CLINICAL TRIAL: NCT00768287
Title: Phase I/II/III Pharmacokinetic and Outcome Study of Recombinant Factor IX Product, IB1001, in Subjects With Hemophilia B
Brief Title: Study of Recombinant Factor IX Product, IB1001, in Subjects With Hemophilia B
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medexus Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IB1001-01
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — IB1001; Factor IX

STUDY DESIGN:
Intervention Model Description: Study Part 1: Randomized, double-blind, cross-over study of pharmacokinetics; Study Part 2: Non-randomized, open-label study of safety and efficacy; Surgical sub-study: Non-randomized, open-label study of safety and efficacy during major surgery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study Part 1 only
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IB1001 (Experimental)
  Interventions: Biological: IB1001
- nonacog alfa (Active Comparator)
  Interventions: Biological: nonacog alfa

INTERVENTIONS:
Biological: IB1001 — Study Part 1: Randomized, double-blind, cross-over study with IB1001 and nonacog alfa; Study Part 2: Non-randomized, open-label evaluation of prophylaxis and on demand IB1001; Surgical Sub-study: Open-label evaluation of IB1001 during major surgery
  Other Names: Recombinant factor IX (rFIX); IXINITY
  Arms: IB1001
Biological: nonacog alfa — Study Part 1: Randomized, double-blind, cross-over study with IB1001 and nonacog alfa
  Other Names: Recombinant factor IX (rFIX); BeneFIX
  Arms: nonacog alfa

SUMMARY:
Primary Objective:

To evaluate the safety (acute effects associated with infusions, and inhibitor development), pharmacokinetics (PK), and efficacy with respect to breakthrough bleeding during prophylaxis and with respect to control of hemorrhaging in both the prophylaxis and on demand groups of IB1001 in subjects with hemophilia B.

Key Secondary Objectives:

To evaluate the ability of IB1001 to provide coverage against bleeding under surgical circumstances; To evaluate the long-term safety and efficacy of IB1001

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be willing to give written Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent, make the required study visits, and follow instructions while enrolled in the study
2. Severe (factor IX activity ≤2 U/dL) hemophilia B subjects on demand therapy with a minimum of 3 bleeding episodes over the preceding 6 months or 6 bleeding episodes over the preceding 12 months; subjects on prophylaxis with a bleeding pattern as above demonstrated prior to starting prophylaxis
3. Immunocompetent (CD4 count >400/mm3) and not receiving immune modulating or chemotherapeutic agents
4. Previously treated patients with a minimum of 150 exposure days to a factor IX preparation
5. Platelet count at least 150,000/mm3
6. Liver function: alanine transaminase [ALT] and aspartate transaminase [AST] ≤2 times the upper limit of the normal range
7. Total bilirubin ≤1.5 times the upper limit of the normal range
8. Renal function: serum creatinine ≤1.25 times the upper limit of the normal range
9. Willingness to participate in the trial for up to 12-15 months
10. European Union (EU), Israel, and Canada: Age of at least 12 years and body weight of ≥40 kilograms to participate in any PK Study or the Surgical Sub-study [the Surgical Sub-study does not apply to the UK]; age of at least 12 years for the prophylaxis and on demand components of the Treatment Phase and Continuation Study

    United States (US): Age of at least 12 years and body weight of ≥40 kilograms to participate in any PK Study or the Surgical Sub-study; age of at least 5 years for the prophylaxis and on demand components of the Treatment Phase and Continuation Study
11. Hemoglobin ≥7 g/dL at the time of the blood draw

Exclusion Criteria:

1. History of factor IX inhibitor ≥0.6 Bethesda units (BU)
2. Existence of another coagulation disorder
3. Evidence of thrombotic disease, fibrinolysis, or disseminated intravascular coagulation (DIC)
4. Use of an investigational drug within 30 days prior to study entry
5. On medications that could impact hemostasis, such as aspirin
6. History of poor compliance, a serious medical or social condition, or any other circumstance that, in the opinion of the investigator, would interfere with participation or compliance with the study protocol
7. History of adverse reaction to either plasma-derived factor IX or recombinant factor IX that interfered with the subject's ability to treat bleeding episodes with a factor IX product

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (10):
  - City of Hope, Duarte, California
  - The Hemophilia Treatment Center of Orthopaedic Hospital, Los Angeles, California
  - Emory University School of Medicine Pediatric Hematology, Atlanta, Georgia
  - Rush University Medical Center-Pediatric Hematology Oncology, Chicago, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - University of Minnesota Center for Bleeding and Clotting Disorder, Minneapolis, Minnesota
  - Hemophilia Treatment Center of Las Vegas, Las Vegas, Nevada
  - Hemophilia and Thrombosis Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas Health Science Center-Houston, Gulf States Hemophilia & Thrombophilia Center, Houston, Texas
- France (2):
  - Centre Regional de Traitement de l 'Hemophilie, Nantes, Loire-Atlantique
  - Hopital Edouard Herriot, Lyon
- India (2):
  - Sahyadri Specialty Hospital, Deccan Gymkhana, Pune, Maharashtra
  - Jehangir Clinical Development Centre, Pune, Maharashtra
- The National Hemophilia Center-Sheba MC, Tel Litwinsky, Ramat Gan, Israel
- Italy (2):
  - Ospedale di Careggi, Florence
  - University of Milan, Milan
- MTZ Clinical Research, Warsaw, Poland
- United Kingdom (5):
  - Royal Free Hospital, London, England
  - Manchester Haemophilia Comprehensive Care Manchester Royal Infirmary, Manchester, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Centre for Haemostasis and Thrombosis, Basingstoke and North Hampshire Foundation Trust, Basingstoke, Hampshire
  - University Hospital of Wales Health Park, Cardiff, Wales

REFERENCES:
- [Result] Collins PW, Quon DVK, Makris M, Chowdary P, Kempton CL, Apte SJ, Ramanan MV, Hay CRM, Drobic B, Hua Y, Babinchak TJ, Gomperts ED. Pharmacokinetics, safety and efficacy of a recombinant factor IX product, trenonacog alfa in previously treated haemophilia B patients. Haemophilia. 2018 Jan;24(1):104-112. doi: 10.1111/hae.13324. Epub 2017 Aug 17. PMID 28833808
- [Derived] Martinowitz U, Shapiro A, Quon DV, Escobar M, Kempton C, Collins PW, Chowdary P, Makris M, Mannucci PM, Morfini M, Valentino LA, Gomperts E, Lee M. Pharmacokinetic properties of IB1001, an investigational recombinant factor IX, in patients with haemophilia B: repeat pharmacokinetic evaluation and sialylation analysis. Haemophilia. 2012 Nov;18(6):881-7. doi: 10.1111/j.1365-2516.2012.02897.x. Epub 2012 Jul 5. PMID 22764744

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects could enter the study at any part and could leave at any time. Of the 77 subjects in the total study population, 32 entered during the PK part, 35 entered during the Treatment part, and 10 entered during the Surgical Substudy. Nine subjects participated only in one Part: 3 only in the PK study and 6 only in the Surgical Substudy
Groups:
- PK: IB1001 First, Then Nonacog Alfa; PK: Nonacog Alfa First, Then IB1001: Pharmacokinetic Study: Randomized, double-blind, cross-over study
- Repeat IB1001 PK: Repeat Pharmacokinetic Study: Non-randomized, open-label study
- IB1001 Prophylaxis; IB1001 On Demand: Treatment Study: Non-randomized, open-label study
- IB1001 Surgical Substudy: Surgical Substudy: Non-randomized, open-label study
Period: Pharmacokinetic Study
Arm/Group | PK: IB1001 First, Then Nonacog Alfa | PK: Nonacog Alfa First, Then IB1001 | Repeat IB1001 PK | IB1001 Prophylaxis | IB1001 On Demand | IB1001 Surgical Substudy
Started | 16 | 16 | 0 | 0 | 0 | 0
Completed | 16 | 16 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Repeat Pharmacokinetic Study
Arm/Group | PK: IB1001 First, Then Nonacog Alfa | PK: Nonacog Alfa First, Then IB1001 | Repeat IB1001 PK | IB1001 Prophylaxis | IB1001 On Demand | IB1001 Surgical Substudy
Started | 0 | 0 | 14 (Eight subjects were part of the IB1001 first group; 6 were from the nonacog alfa first group.) | 0 | 0 | 0
Completed | 0 | 0 | 14 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Study
Arm/Group | PK: IB1001 First, Then Nonacog Alfa | PK: Nonacog Alfa First, Then IB1001 | Repeat IB1001 PK | IB1001 Prophylaxis | IB1001 On Demand | IB1001 Surgical Substudy
Started (29 subjects enrolled from PK study; 4 from Surgery Substudy; 35 directly into Treatment study.) | 0 | 0 | 0 | 58 (1 subject was not assigned a regimen at the start of the study.) | 9 (1 subject was not assigned a regimen at the start of the study.) | 0
Treated | 0 | 0 | 0 | 61 (Subjects could switch treatment regimens. 3 subjects switched from On Demand to Prophylaxis.) | 12 (Subjects could switch treatment regimens. 3 subjects switched from Prophylaxis to On Demand.) | 0
Completed | 0 | 0 | 0 | 58 | 9 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Surgical Sub-study
Arm/Group | PK: IB1001 First, Then Nonacog Alfa | PK: Nonacog Alfa First, Then IB1001 | Repeat IB1001 PK | IB1001 Prophylaxis | IB1001 On Demand | IB1001 Surgical Substudy
Started (Four subjects came from prophylaxis, 3 from on demand, 10 enrolled directly into Surgical Substudy.) | 0 | 0 | 0 | 0 | 0 | 17 (1 female subject was excluded from the efficacy analysis. She was included in the safety population.)
Completed | 0 | 0 | 0 | 0 | 0 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IB1001 Safety Population: Study Population exposed to at least one infusion of IB1001.
Arm/Group | IB1001 Safety Population
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (14.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaska Native | 0
  Race: Asian | 8
  Race: Black or African American | 3
  Race: Caucasian | 61
  Race: Native Hawaiian or Other Pacific Islander | 2
  Race: Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Degree of Hemorrhage Control by Treatment Regimen
Description: Subject rating of bleed control within 6 hours of the time bleeding has stopped:
  1. Excellent: a dramatic response with abrupt pain relief and clear reduction in joint or hemorrhage site size;
  2. Good: pain relief or reduction in hemorrhage site size that may have required an additional infusion for resolution;
  3. Fair: probable or slight beneficial response usually requiring one or more additional infusions for resolution;
  4. Poor: no improvement or condition worsens.
Time Frame: Prophylaxis Group Duration of Treatment: 17.9 ± 9.6 months; On Demand Group Duration of Treatment: 15.9 ± 11.5 months
Population: The 68 patients in the Treatment Study (Part 2) were assigned to an initial treatment regimen as follows: prophylaxis (n=58), on demand (n=9), and unassigned (n=1). Patients were allowed to switch regimens during the course of the study. As a result 61 patients were treated with prophylaxis and 12 patients were treated on demand.
Measure: Count of Units; unit: Bleeding Episodes
Units Other Than Participants: Bleeding Episodes
Groups:
- IB1001 (On Demand): IB1001 50-100 IU/kg at the time of a bleeding episode
- IB1001 (Prophylaxis): IB1001 50-75 IU/kg twice a week
Arm/Group | IB1001 (On Demand) | IB1001 (Prophylaxis)
Number analyzed (Participants) | 12 | 61
Number analyzed (Bleeding Episodes) | 222 | 286
Bleeding Episodes
  Excellent | 53 | 116
  Good | 105 | 74
  Fair | 25 | 28
  Poor | 3 | 9
  Not Rated | 36 | 59

2. Secondary Outcome: Area Under the Curve (0-inf)
Description: Factor IX levels were assessed at the following time points: Pre-infusion, post-infusion at 30 min ± 5 min, 1 hour ± 5 min, 3 hours ± 30 min, 6 hours ± 1 hour, 9 hours ± 1 hour, 12 hours ± 2 hours, 24 hours ± 3 hours, 36 hours ± 3 hours, 48 hours ± 3 hours, 60 hours ± 3 hours, and 72 hours ± 3 hours.
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: IU*hr/dL
Groups:
- IB1001: IB1001 75 ± 5 IU/kg
- Nonacog Alfa: nonacog alfa 75 ± 5 IU/kg
- Repeat IB1001: Repeat PK study of IB1001 75 ± 5 IU/kg 3.1 to 18.6 (median 5.8) months following initial PK study
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
IU*hr/dL | 1572.5 (451.5) | 1656.5 (468.6) | 1530.0 (435.4)

3. Secondary Outcome: Area Under the Curve (0-72 hr)
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: IU*hr/dL
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
IU*hr/dL | 1374.6 (356.4) | 1414.5 (339.4) | 1355.9 (381.2)

4. Secondary Outcome: Terminal Half-life
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
hours | 24.2 (6.9) | 26.4 (13.6) | 24.2 (6.3)

5. Secondary Outcome: Concentration (Max)
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
IU/dL | 73.7 (16.6) | 72.8 (17.5) | 72.7 (15.2)

6. Secondary Outcome: Incremental Recovery
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
IU/dL per IU/kg | 0.98 (0.21) | 0.94 (0.23) | 0.94 (0.18)

7. Secondary Outcome: Mean Residence Time
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
hours | 31.9 (6.4) | 35.4 (13.1) | 30.5 (5.0)

8. Secondary Outcome: Clearance
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: dL/kg*hr
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
dL/kg*hr | 0.051 (0.013) | 0.050 (0.012) | 0.052 (0.015)

9. Secondary Outcome: Volume of Distribution (Steady State)
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | IB1001 | Nonacog Alfa | Repeat IB1001
Number analyzed (Participants) | 32 | 32 | 14
dL/kg | 1.75 (0.57) | 1.81 (0.57) | 1.85 (0.70)

10. Secondary Outcome: Annualized Bleed Rate
Description: Measure was assessed during the Treatment Study
Time Frame: Prophylaxis Group Duration of Treatment: 17.9 ± 9.6 months; On Demand Group Duration of Treatment: 15.9 ± 11.5 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Bleeds/year
Arm/Group | IB1001 (On Demand) | IB1001 (Prophylaxis)
Number analyzed (Participants) | 12 | 61
Bleeds/year | 16.10 [6.6 to 23.7] | 1.52 [0.0 to 3.5]

11. Other Pre Specified Outcome: Blood Loss During Surgery
Description: Surgeon assessment of blood loss during the procedure using the following descriptors: less than expected, expected, or more than expected. Measure was assessed during Surgical Substudy.
Time Frame: During the surgical procedure
Population: Major surgeries include synovectomy, knee or hip replacement, total tooth extraction, surgery for intracranial hemorrhage, radial head excision, arthrodesis, ankle surgery, abdominal surgery, prostatectomy, or surgery for major muscle bleed repair
Measure: Count of Units; unit: Major surgeries
Units Other Than Participants: Major surgeries
Groups:
- IB1001 - Surgical Substudy: IB1001 Bolus Regimen: 120 IU/kg prior to start of procedure, followed by 60 IU/kg 12 hours after the first infusion, and up to 120 IU/kg 24 hours after the first infusion. Bolus infusions continue every 12 hours for a minimum of 3 days; or
  IB1001 Continuous Infusion Regimen: IB1001 infused at a target range of 70% to 110% for a minimum of 3 days post-procedure.
Arm/Group | IB1001 - Surgical Substudy
Number analyzed (Participants) | 16
Number analyzed (Major surgeries) | 19
Major surgeries
  Less than expected | 6
  Expected | 13
  More than expected | 0

12. Other Pre Specified Outcome: Hemostasis Following Surgery
Description: Surgeon assessment of hemostasis at 12 and 24 hours after surgery using the following descriptors: superior, adequate, or poorly controlled. Measure was assessed during Surgical Substudy.
Time Frame: 12 and 24 hours after surgery
Measure: Count of Units; unit: Major surgeries
Units Other Than Participants: Major surgeries
Groups:
- IB1001 (12 Hours) - Surgical Substudy: Hemostasis 12 hours following surgery;
  IB1001 Bolus Regimen: 120 IU/kg prior to start of procedure, followed by 60 IU/kg 12 hours after the first infusion, and up to 120 IU/kg 24 hours after the first infusion. Bolus infusions would continue every 12 hours for a minimum of 3 days; or
  IB1001 Continuous Infusion Regimen: IB1001 infused at a target range of 70% to 110% for a minimum of 3 days post-procedure.
- IB1001 (24 Hours) - Surgical Substudy: Hemostasis 24 hours following surgery;
  IB1001 Bolus Regimen: 120 IU/kg prior to start of procedure, followed by 60 IU/kg 12 hours after the first infusion, and up to 120 IU/kg 24 hours after the first infusion. Bolus infusions would continue every 12 hours for a minimum of 3 days; or
  IB1001 Continuous Infusion Regimen: IB1001 infused at a target range of 70% to 110% for a minimum of 3 days post-procedure.
Arm/Group | IB1001 (12 Hours) - Surgical Substudy | IB1001 (24 Hours) - Surgical Substudy
Number analyzed (Participants) | 16 | 16
Number analyzed (Major surgeries) | 19 | 19
Major surgeries
  Superior | 7 | 7
  Adequate | 12 | 12
  Poorly Controlled | 0 | 0

13. Other Pre Specified Outcome: Number of Surgeries Requiring Blood Transfusions
Description: Measure was assessed during Surgical Substudy.
Time Frame: During the surgical procedure
Measure: Count of Units; unit: Major surgeries
Units Other Than Participants: Major surgeries
Groups:
- IB1001 - Surgical Substudy: IB1001 Bolus Regimen: 120 IU/kg prior to start of procedure, followed by 60 IU/kg 12 hours after the first infusion, and up to 120 IU/kg 24 hours after the first infusion. Bolus infusions would continue every 12 hours for a minimum of 3 days; or
  IB1001 Continuous Infusion Regimen: IB1001 infused at a target range of 70% to 110% for a minimum of 3 days post-procedure.
Arm/Group | IB1001 - Surgical Substudy
Number analyzed (Participants) | 16
Number analyzed (Major surgeries) | 19
Major surgeries
  Blood Transfusion Required | 0
  No Blood Transfusion Required | 19

ADVERSE EVENTS:
Groups:
- IB1001 Safety Population: Adverse Events were only analyzed for the IB1001 safety population; they were not collected per intervention. The safety population is defined as all subjects who received at least one dose of IB1001 in any part of the study.
Arm/Group | IB1001 Safety Population
Serious Adverse Events (participants affected / at risk) | 10/77
Other Adverse Events (participants affected / at risk) | 58/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IB1001 Safety Population (N=77)
Haematoma (Vascular disorders) | 1 (1) — Deemed unrelated to IB1001
Diverticulitis (Infections and infestations) | 1 (3) — Deemed unrelated to IB1001
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) — Deemed unrelated to IB1001
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) — Deemed unrelated to IB1001
Joint injury (Injury, poisoning and procedural complications) | 1 (1) — Deemed unrelated to IB1001
Limb injury (Injury, poisoning and procedural complications) | 1 (1) — Deemed unrelated to IB1001
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Deemed unrelated to IB1001
Mental status changes (Psychiatric disorders) | 1 (1) — Deemed unrelated to IB1001
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) — Deemed unrelated to IB1001
Wound infection (Infections and infestations) | 1 (1) — Deemed unrelated to IB1001
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) — Deemed unrelated to IB1001
Postoperative wound infection (Infections and infestations) | 1 (1) — Deemed unrelated to IB1001
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IB1001 Safety Population (N=77)
Constipation (Gastrointestinal disorders) | 4 (8)
Dairrhoea (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 6 (7)
Pyrexia (General disorders) | 10 (10)
Nasopharyngitis (Infections and infestations) | 9 (18)
Contusion (Injury, poisoning and procedural complications) | 4 (7)
Limb injury (Injury, poisoning and procedural complications) | 8 (8)
Procedural pain (Injury, poisoning and procedural complications) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (10)
Dizziness (Nervous system disorders) | 5 (9)
Headache (Nervous system disorders) | 13 (37)
Insomnia (Psychiatric disorders) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Hypertension (Vascular disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint injury (Injury, poisoning and procedural complications) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No